CLINICAL TRIAL: NCT05492682
Title: A Study to Evaluate the Safety and Immune Activity of PeptiCRAd-1 in Combination With Pembrolizumab in Patients With Injectable Solid Tumors in Indications Known to Express NY-ESO-1 and MAGE-A3
Brief Title: START: Safety and Anti-Tumor Activity of PeptiCRAd-1 in Treatment of Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Valo Therapeutics Oy (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VALO-001; 2021-002529-13 (EudraCT Number)
Record Dates: First submitted 2022-05-18; First posted 2022-08-08 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Melanoma (Skin); Triple-Negative Breast Cancer; Non-Small Cell Lung Cancer; Synovial Sarcoma; Myxoid Liposarcoma; Colorectal Cancer; Osteosarcoma; Sarcoma
MeSH Terms: conditions — Melanoma; Triple Negative Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Sarcoma, Synovial; Liposarcoma, Myxoid; Colorectal Neoplasms; Osteosarcoma; Sarcoma | interventions — Cyclophosphamide; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Patients in Cohort 1 are treated with PeptiCRAd-1 administered i.t.
  Interventions: Drug: PeptiCRAd-1; Drug: Cyclophosphamide; Drug: Pembrolizumab
- Cohort 2 (Experimental): Patients in Cohort 2 are treated with PeptiCRAd-1 administered i.t. and s.c.
  Interventions: Drug: PeptiCRAd-1; Drug: Cyclophosphamide; Drug: Pembrolizumab

INTERVENTIONS:
Drug: PeptiCRAd-1 — All patients will receive PeptiCRAd-1.
Drug: Cyclophosphamide — All patients will be pre-treated with one single dose of Cyclophosphamide.
Drug: Pembrolizumab — All patients will receive 6 doses of Pembrolizumab within the study.

SUMMARY:
This study is being conducted to explore the immunological mechanism of action of Peptide-coated Conditionally Replicating Adenovirus-1 (PeptiCRAd-1) plus Checkpoint inhibitor (CPI) therapy in multiple cancer types, as well as to obtain early information on the safety of this combination therapy.

DETAILED DESCRIPTION:
This is a Phase I, open-label, non-randomized, first-in-human study. All patients will be pre-treated with a low dose of intravenous (i.v.) Cyclophosphamide (CPO) followed by monotherapy doses of PeptiCRAd-1. PeptiCRAd-1 will be administered by intratumoral (i.t.) injection (Cohort 1) and by i.t. and subcutaneous (s.c.) injection (Cohort 2) followed by combination therapy with PeptiCRAd-1 and i.v. CPI (pembrolizumab).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Male or female, ≥18 years of age.
3. Patients with any 1 of the following histologically confirmed tumors and who qualifies for new or continued CPI therapy and relapsing to/after standard therapy or the patient has refused or does not tolerate standard therapy:

   * Inoperable/metastatic cutaneous malignant melanoma
   * Relapsed or newly diagnosed locally advanced inoperable/metastatic TNBC
   * Inoperable advanced/metastatic non-squamous NSCLC
   * Inoperable and/or advanced Synovial or myxoid round cell sarcoma
   * Inoperable and/or advanced osteosarcoma
   * Inoperable and/or advanced colorectal cancer, patients assessed as positive for NY-ESO-1 or MAGE-A3 expression at baseline
   * Inoperable and/or advanced/metastatic sarcoma, patients assessed as positive for NY-ESO-1 or MAGE-A3 expression at baseline
4. Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
5. Tumor lesion which is deemed feasible for biopsy and injection
6. ECOG/WHO performance status 0 to 1.
7. Acceptable liver and renal function, defined as:

   * Total bilirubin ≤1.5 x upper limit of normal (ULN; does not include patients with Gilbert's Disease), and
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3.0 x ULN, and
   * Serum creatinine ≤1.5 x ULN
8. Acceptable hematological function, defined as:

   * Hemoglobin ≥9 g/dL, and
   * Neutrophils ≥1.5 x 109/L, and
   * Platelet count ≥100 x 109/L Patients may be transfused to meet the hemoglobin entry criteria.
9. Acceptable coagulation status defined by international normalized ratio (INR) of blood clotting, prothrombin time and activated partial thromboplastin time within ≤1.5 x upper limit of normal.
10. Negative pregnancy test at screening in all women of childbearing potential (WOCBP). Such patients must agree to use a highly effective method of contraception (Appendix 1) during study intervention and for 3 months after the last virus treatment, 4 months after the last dose of pembrolizumab, and 12 months after CPO dosing. Male patients and male partners of female patients must also use barrier contraception, i.e., condom, for the time periods specified for WOCBP, plus a further 3 month period.

    Urine pregnancy tests should have a sensitivity of at least 25 mIU/mL for human chorionic gonadotropin (hCG). If the urine test is positive, it must be followed by a quantitative analysis of hCG concentration in blood.
11. Prior therapy with an immune CPI is allowed provided a 6-week washout period is observed for patients with prior programmed cell death (PD)1 or PDL1 treatment

Exclusion Criteria:

1. Receipt of any oncolytic virus treatment, or administration of a vaccine containing live virus within 4 weeks before Day 1.
2. Use of significant immunosuppressive medication, including high dose corticosteroid (defined as the equivalent of >10 mg/day prednisone) within 4 weeks before Day 1. Inhaled or topical corticosteroid use is allowed.
3. Prior or concomitant radiotherapy within 4 weeks before Day 1.
4. Participation in a study with an investigational drug or device within 4 weeks prior to Day 1.
5. Active bacterial, viral, or fungal infection that requires systemic therapy.
6. Active autoimmune disease that has required systemic treatment in the past two years.
7. Concomitant disease or condition that could interfere with the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the patient, if included in this study.
8. Any concomitant medical condition requiring receipt of a therapeutic anticoagulant that, in the opinion of the treating physician, cannot safely be withheld to allow for repeated injection of PeptiCRAd 1 and tumor biopsies.
9. Known infection with human immunodeficiency virus, hepatitis B, or hepatitis C or active tuberculosis.
10. Known active central nervous system metastases. Patients with leptomeningeal disease, carcinomatous meningitis, symptomatic brain metastases, or radiographic signs of CNS hemorrhage are excluded.

    Note: Participants with asymptomatic brain metastases (i.e. off corticosteroids and anticonvulsants for at least 7 days) are permitted.
11. Any prior severe AE according to Common Terminology Criteria for Adverse Events (CTCAE), severe hypersensitivity reaction attributed to prior anti-PD1 or PDL1 therapy or components of the study intervention or has a history of any contraindication that, in the investigator's opinion, would contraindicate pembrolizumab administration such as:

    * Resolution of side effect of prior anti-PD1 or PDL1 therapy to Grade 1
    * Grade 2 or higher pneumonitis
    * Grade 4 AST or ALT elevation
    * Grade 3 or higher colitis attributable to immunotherapy Note: in the absence of clinical symptoms of pancreatitis, elevations of amylase or lipase are not contraindications to therapy on this trial.
12. History of or planned tissue / organ transplant.
13. Females who are pregnant or breast feeding or expecting to conceive within the projected duration of the study starting with the screening visit or males expecting to father children within the projected duration of the study starting with the screening visit.
14. Unwillingness or inability to comply with the study protocol for any reason.
15. Admission to an institution by virtue of an order issued by the judicial or administrative authorities.
16. Sponsor or Contract Research Organization employees, or employees under the direct supervision of the investigator or the investigational sites and/or involved directly in the study.
17. Prior or concurrent malignancy, unless the natural history or treatment of the disease does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-02-02 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Measurement of Safety and tolerability indexes (Incidence of TEAEs, SAEs and DLTs as assessed by CTCAE version 5.0 and changes in assessed safety parameters) for PeptiCRAd-1 monotherapy. | From study protocol day 1 (baseline) until 1 month
  The incidence and characteristics of treatment-emergent adverse events (TEAEs), serious adverse events (SAEs) and dose-limiting toxicities (DLTs) will be assessed by CTCAE version 5.0 and changes from baseline in assessed safety parameters (Hematology tests, Clinical Chemistry safety tests, urine analysis ECOG/WHO performance status, vital signs) are measured in patients receiving PeptiCRAd-1 monotherapy in order to evaluate the safety and tolerability.
Measurement of Safety and tolerability indexes (Incidence of TEAEs, SAEs and DLTs as assessed by CTCAE version 5.0 and changes in assessed safety parameters) for PeptiCRAd-1 and CPI combination. | From first month through study completion, an average of 4.5 months.
  The incidence and characteristics of TEAEs, SAEs and DLTs will be assessed by CTCAE version 5.0 and changes from baseline in assessed safety parameters (Hematology tests, Clinical Chemistry safety tests, urine analysis ECOG/WHO performance status, vital signs) are measured in patients receiving PeptiCRAd-1 and CPI combination in order to evaluate the safety and tolerability.

SECONDARY OUTCOMES:
Measurement of New York Esophageal Squamous Cell Carcinoma-1 (NY-ESO-1) and Melanoma-associated antigen 3 (MAGE A3) specific T-cells in peripheral blood. | Change from Baseline through study completion, an average of 5 months.
  Presence vs. no presence of cellular immune response.
Measurement of NY-ESO-1 and MAGE A3 antibodies in serum. | Change from Baseline to an average of 3,5 months
  Presence vs. no presence of humoral response.
To determine the number of tumor infiltrating lymphocytes (TILs) in tumor mass. | Change from Baseline to an average of 3 months
  Number of TILs in tumor biopsies.
To determine objective response rate (ORR). | Change from Baseline through study completion, an average of 5 months.
  Objective responses according to RECIST 1.1, iRECIST, itRECIST and PERCIST 1.0.
To determine overall survival. | Change from Baseline through study completion, an average of 5 months.
  Overall survival presented in Kaplan-Meier plot.
Correlation between immune activation in peripheral blood and tumor mass and clinical outcome. | Change from Baseline through study completion, an average of 5 months.
  Correlation between immune activation (immunological variables) in peripheral blood and tumor mass and clinical outcome (ORR, OS).

OTHER OUTCOMES:
Measurement of PFS according to RECIST 1.1, itRECIST, and PERCIST 1.0. | Change from Baseline through study completion, an average of 5 months.
  Progression free survival (PFS) is measured, according to RECIST 1.1, iRECIST, itRECIST, and PERCIST 1.0, and will be presented using the Kaplan-Meier approach.
Measurement of virus shedding profiles (presence of infective virus and virus DNA in blood, urine, buccal, fecal and injection site swabs by infectivity assay and qPCR). | Changes from baseline to an average of 3,5 months.
  Presence of infective virus (infectivity assay) and virus DNA (quantitative polymerase chain reaction, qPCR) will be measured in blood, urine, buccal, fecal and injection site swabs.
Immune phenotyping in tumor mass. | Changes from baseline to to an average of 3 months
  Measurement of biological and immunological changes (including number of T-cells) in biopsies of injected and non-injected tumors over time.
Measurement of the phenotype of circulating immune cells in peripheral blood. | Change from Baseline through study completion, an average of 5 months.
  The immunological landscape in peripheral blood will be determined.

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - Krankenhaus Nordwest, Frankfurt
  - National Center for Tumor Diseases, Heidelberg
  - Universitätsklinikum Tübingen, Tübingen